CLINICAL TRIAL: NCT02611778
Title: Efficacy and Safety of the Biosimilar Ranibizumab FYB201 in Comparison to Lucentis in Patients With Neovascular Age-related Macular Degeneration
Acronym: COLUMBUS-AMD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bioeq GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FYB201-C2015-01-P3
Record Dates: First submitted 2015-11-19; First posted 2015-11-23 (Estimated); Results first posted 2021-09-30 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Age-related Macular Degeneration (AMD)
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FYB201 (Experimental): FYB201 is provided as single use vials and will be administered by intra-vitreal injection.
  Interventions: Biological: ranibizumab
- Lucentis (Active Comparator): Lucentis® is provided as single use vials and will be administered by intra-vitreal injection.
  Interventions: Biological: ranibizumab

INTERVENTIONS:
Biological: ranibizumab

SUMMARY:
The purpose of this study is to determine the efficacy and safety of the biosimilar ranibizumab FYB201 in comparison to Lucentis in patients with neovascular age-related macular degeneration.

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 50 years of either gender
* Signed informed consent form must be obtained before any study-related procedure is performed
* Willingness and ability to undertake all scheduled visits and assessments
* Women must be postmenopausal or surgically sterile
* Newly diagnosed, angiographically documented, primary active Choroidal Neovascularization (CNV) lesion secondary to age-related macular degeneration (AMD)
* Sufficiently clear ocular media and adequate pupillary dilation to permit good quality ocular imaging
* Best-corrected Visual Acuity (BCVA) in the study eye, determined by standardized Early Treatment Diabetic Retinopathy Study (ETDRS) testing, between 20/32 (0.63) and 20/100 (0.2) Snellen equivalent
* Foveal Center Point (FCP) retinal thickness in at Screening ≥ 350 µm
* BCVA in the fellow eye, determined by standardized ETDRS testing, at least 20/100 (0.2) Snellen equivalent

Exclusion criteria:

* Employees of clinical study sites, individuals directly involved with the conduct of the study or immediate family members thereof, prisoners, and persons who are legally institutionalized
* Any previous treatment with intravitreal (IVT) anti-vascular endothelial growth factor (VEGF) agent in either eye
* History of vitrectomy, macular surgery or other surgical intervention for AMD in the study eye
* History of IVT or periocular injections of corticosteroids or device implantation within six months prior to Screening in the study eye
* Prior treatment with verteporfin (photodynamic therapy), transpupillary thermotherapy, radiation therapy, or retinal laser treatment (e.g. focal laser photocoagulation) in the study eye
* Topical ocular corticosteroids administered for at least 30 consecutive days within three months prior to Screening
* Any other intraocular surgery (including cataract surgery) in the study eye within three months prior to Screening
* Sub- or intra-retinal hemorrhage that comprises more than 50% of the entire lesion in the study eye
* Fibrosis or atrophy involving the center of the fovea or influencing central visual function in the study eye
* CNV in either eye due to other causes, such as ocular histoplasmosis, trauma, or pathologic myopia
* Retinal pigment epithelial tear involving the macula in the study eye
* History of full-thickness macular hole in the study eye
* History of retinal detachment in the study eye
* Current vitreous hemorrhage in the study eye
* Spherical equivalent of the refractive error in the study eye demonstrating more than 8 diopters of myopia
* For patients who have undergone prior refractive or cataract surgery in the study eye, the preoperative refractive error in the study eye cannot exceed 8 diopters of myopia
* History of corneal transplant in the study eye
* Aphakia in the study eye. Absence of an intact posterior capsule is allowed if it occurred as a result of Yttrium-Aluminium-Garnet (YAG) laser posterior capsulotomy in association with prior posterior chamber intraocular lens (IOL) implantation
* Active or recent (within 4 weeks) intraocular inflammation of clinical significance in the study eye such as active infections of the anterior segment (excluding mild blepharitis) including conjunctivitis, keratitis, scleritis, uveitis or endophthalmitis
* Uncontrolled hypertension or glaucoma in the study eye (defined as intraocular pressure (IOP) ≥30 mm Hg, despite treatment with anti-glaucomatous medication)
* Ocular disorders in the study eye (i.e. retinal detachment, pre-retinal membrane of the macula or cataract with significant impact on visual acuity) at the time of enrollment that may confound interpretation of study results and compromise visual acuity
* Any concurrent intraocular condition in the study eye (e.g. glaucoma, cataract or diabetic retinopathy) that, in the opinion of the Investigator, would either require surgical intervention during the study to prevent or treat visual loss that might result from that condition or affect interpretation of study results.
* Use of other investigational drugs (excluding vitamins, minerals) within 30 days or 5 half-lives from Screening, whichever is longer
* Any type of advanced, severe or unstable disease, including any medical condition (controlled or uncontrolled) that could be expected to progress, recur, or change to such an extent that it may bias the assessment of the clinical status of the patient to a significant degree or put the patient at special risk
* Stroke or myocardial infarction within three months prior to Screening
* Presence of uncontrolled systolic blood pressure > 160 mmHg or uncontrolled diastolic blood pressure > 100 mmHg
* Known hypersensitivity to the investigational drug (ranibizumab or any component of the ranibizumab formulation) or to drugs of similar chemical class or to fluorescein or any other component of fluorescein formulation
* Current or planned use of systemic medications known to be toxic to the lens, retina or optic nerve, including deferoxamine, chloroquine/hydroxychloroquine (Plaquenil®), tamoxifen, phenothiazines and ethambutol
* History of recurrent significant infections and/or current treatment for active systemic infection
* Pregnancy or lactation
* Systemic treatment with high doses of corticosteroids (administration of >10 mg/day of prednisolone equivalent) during the last six months prior to Screening
* Inability to comply with study or follow-up procedures
* Any diagnosis and/or signs of nAMD requiring treatment with an IVT anti-VEGF agent (e.g. aflibercept, bevacizumab, ranibizumab) within the screening period or at study treatment initiation (Visit 1) in the fellow eye

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 712 (Actual)
Dates: Start 2015-12-19 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank G. Holz, Prof. Dr., Principal Investigator — University of Bonn, Department of Ophthalmology
Locations (58):
- Research Site, Vienna, Austria
- Czechia (5):
  - Research Site, Brno
  - Research Site, Ostrava
  - Research Site, Pilsen
  - Research Site, Prague
  - Research Site, Zlín
- France (4):
  - Research Site, Dijon
  - Research Site, Lyon
  - Research Site, Nantes
  - Research Site, Paris
- Germany (8):
  - University of Bonn, Department of Ophthalmology, Bonn
  - Research Site, Dresden
  - Research Site, Freiburg im Breisgau
  - Research Site, Göttingen
  - Research Site, Hanover
  - Research Site, Leipzig
  - Research Site, Mainz
  - Research Site, Tübingen
- Hungary (6):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Nyíregyháza
  - Research Site, Pécs
  - Research Site, Szeged
  - Research Site, Zalaegerszeg
- Israel (9):
  - Research Site, Beersheba
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
  - Research Site, Rehovot
  - Research Site, Tel Aviv
  - Research Site, Zrifin
- Italy (6):
  - Research Site, Bologna
  - Research Site, Chieti
  - Research Site, Milan
  - Research Site, Pisa
  - Research Site, Roma
  - Research Site, Torino
- Poland (6):
  - Research Site, Bydgoszcz
  - Research Site, Lodz
  - Research Site, Rzeszów
  - Research Site, Tarnowskie Góry
  - Research Site, Tarnów
  - Research Site, Warsaw
- Russia (3):
  - Research Site, Kazan'
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- Spain (3):
  - Research Site, Barcelona
  - Research Site, Valencia
  - Research Site, Zaragoza
- Ukraine (2):
  - Research Site, Kyiv
  - Research Site, Odesa
- United Kingdom (5):
  - Research Site, Bradford
  - Research Site, Bristol
  - Research Site, Camberley
  - Research Site, London
  - Research Site, Rugby

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All 712 patients were screened for eligibility before participating in the active treatment phase of the study, resulting in 722 screenings due to 10 rescreenings. Subjects were not to be entered to trial treatment if any of the eligibility criteria were violated. Of the 712 distinct patients, 477 patients were randomized and treated.
Groups:
- FYB201: Patients received FYB201 at a dose of 0.5mg (0.05mL of a 10mg/mL solution) as twelve monthly intravitreal injections
- Lucentis: Patients received Lucentis (ranibizumab) at a dose of 0.5mg (0.05mL of a 10mg/mL solution) as twelve monthly intravitreal injections
Period: Overall Study
Arm/Group | FYB201 | Lucentis
Started | 238 | 239
Completed | 226 | 226
Not Completed | 12 | 13
Not completed — Withdrawal by Subject | 2 | 8
Not completed — Adverse Event | 1 | 2
Not completed — Death | 2 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 3 | 1
Not completed — Need for alternative treatment | 1 | 0
Not completed — Other Reason | 2 | 1

BASELINE CHARACTERISTICS:
Population: Safety Set (SAF): The safety set comprised all patients who had received at least one injection with investigational medicinal product.
Groups:
- Total: Total of all reporting groups
Arm/Group | FYB201 | Lucentis | Total
Number analyzed (Participants) | 238 | 239 | 477
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.9 (8.26) | 76.1 (7.84) | 75.5 (8.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135 | 134 | 269
  Male | 103 | 105 | 208
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 236 | 233 | 469
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) [Letters] After 8 Weeks
Description: The primary endpoint was the absolute change from baseline in BCVA by Early Treatment Diabetic Retinopathy Study (ETDRS) letters after 2 months (8 weeks) of treatment.
Time Frame: Baseline and Week 8
Population: FAS_US: The FAS_US was based on the intention to treat principle (i.e., patients were analyzed according to their randomized treatment irrespective of the treatment they actually received) and included all patients who received at least one injection of IMP, and for whom BCVA results at least after 1 month were available and who had a screening BCVA between 20/32 and 20/100 Snellen equivalent in the study eye.
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | FYB201 | Lucentis | Total
Number analyzed (Participants) | 228 | 233 | 475
letters | 5.1 (7.52) | 5.6 (8.63) | 5.4 (8.10)
Statistical Analysis 1: Comparison: FYB201 vs Lucentis; The hypothesis of biosimilarity of FYB201 and Lucentis was tested with a two-sided equivalence test with an equivalence margin of 3 ETDRS letters. An ANCOVA model was used with the change in BCVA between baseline and Week 8 as the dependent variable, the baseline BCVA as covariate, and the country and the treatment group as fixed effects; Test type: Equivalence — The confidence interval (CI) for treatment difference (FYB201 - Lucentis) was calculated using Least Square Means. If the 90% CI was completely contained in the interval ]-3.5;3.5[ ETDRS letters, equivalence of FYB201 and Lucentis could be concluded; ANCOVA; Difference in least square means = -0.4, 90% CI 2-sided [-1.6 to 0.9], Standard Error of Mean 0.76 — An ANCOVA model was used for the analysis with the change in BCVA between baseline and Week 8 as the dependent variable, the baseline BCVA as covariate, and (pooled) country and treatment group as fixed effects

2. Secondary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) [Letters] After 24 Weeks
Description: Absolute change from baseline in BCVA by Early Treatment Diabetic Retinopathy Study (ETDRS) letters after 24 weeks of treatment.
Time Frame: Baseline and Week 24
Population: FAS_US
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | FYB201 | Lucentis | Total
Number analyzed (Participants) | 230 | 232 | 462
letters | 6.9 (10.12) | 7.1 (10.42) | 7.0 (10.26)
Statistical Analysis 1: Comparison: FYB201 vs Lucentis; There was no formal hypothesis testing; Test type: Other; ANCOVA; Difference in least square means = -0.0, 90% CI 2-sided [-1.6 to 1.5], Standard Error of Mean 0.96 — An ANCOVA model was used for the analysis with the change in BCVA between baseline and Week 24 as the dependent variable, the baseline BCVA as covariate, and (pooled) country and treatment group as fixed effects

3. Secondary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) [Letters] After 48 Weeks
Description: Absolute change from baseline in BCVA by Early Treatment Diabetic Retinopathy Study (ETDRS) letters after 48 weeks of treatment.
Time Frame: Baseline and Week 48
Population: FAS_US
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | FYB201 | Lucentis | Total
Number analyzed (Participants) | 225 | 225 | 450
letters | 7.8 (11.67) | 8.0 (11.31) | 7.9 (11.48)
Statistical Analysis 1: Comparison: FYB201 vs Lucentis; There was no formal hypothesis testing; Test type: Other; ANCOVA; Difference in least square means = -0.1, 90% CI 2-sided [-1.8 to 1.7], Standard Error of Mean 1.08 — An ANCOVA model was used for the analysis with the change in BCVA between baseline and Week 48 as the dependent variable, the baseline BCVA as covariate, and (pooled) country and treatment group as fixed effects

4. Secondary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) [Letters] After 12 Months
Description: Absolute change from baseline in BCVA by Early Treatment Diabetic Retinopathy Study (ETDRS) letters after 12 months, calculated as the average of the changes from baseline to Week 40, to Week 44 and to Week 48.
Time Frame: Baseline and 12 Months
Population: FAS_US
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | FYB201 | Lucentis | Total
Number analyzed (Participants) | 228 | 227 | 455
letters | 7.8 (11.19) | 7.9 (11.01) | 7.8 (11.09)
Statistical Analysis 1: Comparison: FYB201 vs Lucentis; There was no formal hypothesis testing; Test type: Other; ANCOVA; Difference in least square means = 0.1, 90% CI 2-sided [-1.6 to 1.8], Standard Error of Mean 1.04 — An ANCOVA model was used for the analysis with the change in BCVA between baseline and 12 months (average of Weeks 40, 44 and 48) as the dependent variable, the baseline BCVA as covariate, and (pooled) country and treatment group as fixed effects

5. Secondary Outcome: Change in Foveal Centre Point (FCP) Retinal Thickness From Baseline to Week 24
Description: Absolute change in Foveal Centre Point (FCP) retinal thickness [µm] from baseline to Week 24
Time Frame: Baseline and Week 24
Population: FAS_US
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | FYB201 | Lucentis | Total
Number analyzed (Participants) | 218 | 221 | 439
µm | -203.94 (147.104) | -205.45 (147.199) | -204.70 (146.986)
Statistical Analysis 1: Comparison: FYB201 vs Lucentis; There was no formal hypothesis testing; Test type: Other; ANCOVA; Difference in least square means = 0.69, 90% CI 2-sided [-18.22 to 19.60], Standard Error of Mean 11.469 — An ANCOVA model was used for the analysis with the change in FCP retinal thickness between baseline and Week 24 as the dependent variable, the baseline FCP retinal thickness as covariate, and (pooled) country and treatment group as fixed effects

6. Secondary Outcome: Change in Foveal Centre Point (FCP) Retinal Thickness From Baseline to Week 48
Description: Absolute change in Foveal Centre Point (FCP) retinal thickness [µm] from baseline to Week 48
Time Frame: Baseline and Week 48
Population: FAS_US
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | FYB201 | Lucentis | Total
Number analyzed (Participants) | 219 | 220 | 439
µm | -213.26 (161.323) | -211.02 (151.950) | -212.14 (156.521)
Statistical Analysis 1: Comparison: FYB201 vs Lucentis; There was no formal hypothesis testing; Test type: Other; ANCOVA; Difference in least square means = 2.68, 90% CI 2-sided [-16.49 to 21.85], Standard Error of Mean 11.632 — An ANCOVA model was used for the analysis with the change in FCP retinal thickness between baseline and Week 48 as the dependent variable, the baseline FCP retinal thickness as covariate, and (pooled) country and treatment group as fixed effects

7. Secondary Outcome: Change in Foveal Central Subfield (FCS) Retinal Thickness From Baseline to Week 24
Description: Absolute change in Foveal Central Subfield (FCS) retinal thickness [µm] from baseline to Week 24
Time Frame: Baseline and Week 24
Population: FAS_US
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | FYB201 | Lucentis | Total
Number analyzed (Participants) | 211 | 220 | 431
µm | -180.37 (128.522) | -181.63 (126.466) | -181.02 (127.330)
Statistical Analysis 1: Comparison: FYB201 vs Lucentis; There was no formal hypothesis testing; Test type: Other; ANCOVA; Difference in least square means = -5.91, 90% CI 2-sided [-22.62 to 10.80], Standard Error of Mean 10.136 — An ANCOVA model was used for the analysis with the change in FCS retinal thickness between baseline and Week 24 as the dependent variable, the baseline FCS retinal thickness as covariate, and (pooled) country and treatment group as fixed effects

8. Secondary Outcome: Change in Foveal Central Subfield (FCS) Retinal Thickness From Baseline to Week 48
Description: Absolute change in Foveal Central Subfield (FCS) retinal thickness [µm] from baseline to Week 48
Time Frame: Baseline and Week 48
Population: FAS_US
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | FYB201 | Lucentis | Total
Number analyzed (Participants) | 207 | 213 | 420
µm | -182.85 (134.588) | -190.75 (128.691) | -186.86 (131.532)
Statistical Analysis 1: Comparison: FYB201 vs Lucentis; There was no formal hypothesis testing; Test type: Other; ANCOVA; Difference in least square means = 3.68, 90% CI 2-sided [-13.28 to 20.63], Standard Error of Mean 10.285 — An ANCOVA model was used for the analysis with the change in FCS retinal thickness between baseline and Week 48 as the dependent variable, the baseline FCS retinal thickness as covariate, and (pooled) country and treatment group as fixed effects

9. Secondary Outcome: Change in Total Lesion Area From Baseline to Week 24
Description: Absolute change in total lesion area [mm²] from baseline to Week 24
Time Frame: Baseline and Week 24
Population: FAS_US
Measure: Mean (Standard Deviation); unit: mm²
Arm/Group | FYB201 | Lucentis | Total
Number analyzed (Participants) | 213 | 207 | 420
mm² | -0.5742 (4.79222) | -0.7113 (5.35854) | -0.6418 (5.07361)
Statistical Analysis 1: Comparison: FYB201 vs Lucentis; There was no formal hypothesis testing; Test type: Other; ANCOVA; Difference in least square means = 0.070, 90% CI 2-sided [-0.706 to 0.846], Standard Error of Mean 0.4709 — An ANCOVA model was used for the analysis with the change in total lesion area between baseline and Week 24 as the dependent variable, the baseline total lesion area as covariate, and (pooled) country and treatment group as fixed effects

10. Secondary Outcome: Change in Total Lesion Area From Baseline to Week 48
Description: Absolute change in total lesion area [mm²] from baseline to Week 48
Time Frame: Baseline and Week 48
Population: FAS_US
Measure: Mean (Standard Deviation); unit: mm²
Arm/Group | FYB201 | Lucentis | Total
Number analyzed (Participants) | 163 | 166 | 329
mm² | -0.6382 (4.81194) | -1.1814 (5.42770) | -0.9123 (5.13128)
Statistical Analysis 1: Comparison: FYB201 vs Lucentis; There was no formal hypothesis testing; Test type: Other; ANCOVA; Difference in least square means = 0.342, 90% CI 2-sided [-0.547 to 1.230], Standard Error of Mean 0.5387 — An ANCOVA model was used for the analysis with the change in total lesion area between baseline and Week 48 as the dependent variable, the baseline total lesion area as covariate, and (pooled) country and treatment group as fixed effects

11. Secondary Outcome: Change in NEI VFQ-25 Composite Score From Baseline to Week 24
Description: Absolute change from baseline to Week 24 in vision-related functioning and well-being measured by the National Eye Institute Visual Function Questionnaire 25 (NEI VFQ-25) composite score.
  The NEI VFQ-25 is a 25 question quality of life questionnaire with possible item scores between 0 and 100. Higher scores represent better functioning. The composite score is calculated as average over all non-missing item scores.
Time Frame: Baseline and Week 24
Population: FAS_US
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FYB201 | Lucentis | Total
Number analyzed (Participants) | 228 | 230 | 458
score on a scale | 3.59 (9.632) | 3.55 (11.237) | 3.57 (10.457)
Statistical Analysis 1: Comparison: FYB201 vs Lucentis; There was no formal hypothesis testing; Test type: Other; ANCOVA; Difference in least square means = 0.21, 90% CI 2-sided [-1.25 to 1.67], Standard Error of Mean 0.886 — An ANCOVA model was used for the analysis with change in NEI VFQ-25 composite score between baseline and Week 24 as dependent variable, baseline NEI VFQ-25 composite score as covariate, and (pooled) country and treatment group as fixed effects

12. Secondary Outcome: Change in NEI VFQ-25 Composite Score From Baseline to Week 48
Description: Absolute change from baseline to Week 48 in vision-related functioning and well-being measured by the National Eye Institute Visual Function Questionnaire 25 (NEI VFQ-25) composite score.
  The NEI VFQ-25 is a 25 question quality of life questionnaire with possible item scores between 0 and 100. Higher scores represent better functioning. The composite score is calculated as average over all non-missing item scores.
Time Frame: Baseline and Week 48
Population: FAS_US
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FYB201 | Lucentis | Total
Number analyzed (Participants) | 224 | 222 | 446
score on a scale | 5.30 (12.205) | 3.75 (13.190) | 4.53 (12.714)
Statistical Analysis 1: Comparison: FYB201 vs Lucentis; There was no formal hypothesis testing; Test type: Other; ANCOVA; Difference in least square means = 1.73, 90% CI 2-sided [0.04 to 3.42], Standard Error of Mean 1.027 — An ANCOVA model was used for the analysis with change in NEI VFQ-25 composite score between baseline and Week 48 as dependent variable, baseline NEI VFQ-25 composite score as covariate, and (pooled) country and treatment group as fixed effects

13. Secondary Outcome: Active CNV Leakage at Week 24
Description: Number and percentage of patients with active CNV leakage at Week 24
Time Frame: Baseline and Week 24
Population: FAS_US
Measure: Count of Participants; unit: Participants
Arm/Group | FYB201 | Lucentis | Total
Number analyzed (Participants) | 221 | 219 | 440
Participants
  CNV leakage | 115 | 111 | 226
  No CNV leakage | 106 | 108 | 214

14. Secondary Outcome: Active CNV Leakage at Week 48
Description: Number and percentage of patients with active CNV leakage at Week 48
Time Frame: Baseline and Week 48
Population: FAS_US
Measure: Count of Participants; unit: Participants
Arm/Group | FYB201 | Lucentis | Total
Number analyzed (Participants) | 211 | 196 | 407
Participants
  CNV leakage | 119 | 115 | 234
  No CNV leakage | 92 | 81 | 173

15. Secondary Outcome: Fluid-free Macula at Each Visit
Description: Number and percentage of patients with fluid-free macula at each visit
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48
Population: FAS_US
Measure: Count of Participants; unit: Participants
Arm/Group | FYB201 | Lucentis | Total
Number analyzed (Participants) | 237 | 238 | 475
Participants
  Baseline: number analyzed (Participants) | 236 | 236 | 472
  Baseline: Fluid-free macula | 0 | 2 | 2
  Baseline: No fluid-free macula | 236 | 234 | 470
  Week 4: number analyzed (Participants) | 230 | 226 | 456
  Week 4: Fluid-free macula | 43 | 38 | 81
  Week 4: No fluid-free macula | 187 | 188 | 375
  Week 8: number analyzed (Participants) | 223 | 230 | 453
  Week 8: Fluid-free macula | 69 | 62 | 131
  Week 8: No fluid-free macula | 154 | 168 | 322
  Week 12: number analyzed (Participants) | 227 | 231 | 458
  Week 12: Fluid-free macula | 86 | 76 | 162
  Week 12: No fluid-free macula | 141 | 155 | 296
  Week 16: number analyzed (Participants) | 223 | 236 | 459
  Week 16: Fluid-free macula | 87 | 87 | 174
  Week 16: No fluid-free macula | 136 | 149 | 285
  Week 20: number analyzed (Participants) | 226 | 234 | 460
  Week 20: Fluid-free macula | 80 | 97 | 177
  Week 20: No fluid-free macula | 146 | 137 | 283
  Week 24: number analyzed (Participants) | 227 | 231 | 458
  Week 24: Fluid-free macula | 86 | 100 | 186
  Week 24: No fluid-free macula | 141 | 131 | 272
  Week 28: number analyzed (Participants) | 226 | 219 | 445
  Week 28: Fluid-free macula | 86 | 98 | 184
  Week 28: No fluid-free macula | 140 | 121 | 261
  Week 32: number analyzed (Participants) | 222 | 221 | 443
  Week 32: Fluid-free macula | 91 | 96 | 187
  Week 32: No fluid-free macula | 131 | 125 | 256
  Week 36: number analyzed (Participants) | 225 | 218 | 443
  Week 36: Fluid-free macula | 83 | 99 | 182
  Week 36: No fluid-free macula | 142 | 119 | 261
  Week 40: number analyzed (Participants) | 220 | 217 | 437
  Week 40: Fluid-free macula | 87 | 102 | 189
  Week 40: No fluid-free macula | 133 | 115 | 248
  Week 44: number analyzed (Participants) | 221 | 220 | 441
  Week 44: Fluid-free macula | 92 | 104 | 196
  Week 44: No fluid-free macula | 129 | 116 | 245
  Week 48: number analyzed (Participants) | 225 | 221 | 446
  Week 48: Fluid-free macula | 105 | 108 | 213
  Week 48: No fluid-free macula | 120 | 113 | 233

16. Secondary Outcome: Anti-drug Antibodies by Scheduled eCRF Visit
Description: Frequency of patients with anti-drug antibodies (ADAs) by scheduled eCRF visit
Time Frame: Baseline and Weeks 1, 4, 12, 24, 48
Population: SAF
Measure: Count of Participants; unit: Participants
Arm/Group | FYB201 | Lucentis | Total
Number analyzed (Participants) | 238 | 239 | 477
Participants
  Baseline: number analyzed (Participants) | 234 | 238 | 472
  Baseline: Positive anti-drug antibodies | 0 | 5 | 5
  Baseline: Negative anti-drug antibodies | 234 | 233 | 467
  Week 1: number analyzed (Participants) | 28 | 29 | 57
  Week 1: Positive anti-drug antibodies | 0 | 0 | 0
  Week 1: Negative anti-drug antibodies | 28 | 29 | 57
  Week 4: number analyzed (Participants) | 226 | 228 | 454
  Week 4: Positive anti-drug antibodies | 2 | 2 | 4
  Week 4: Negative anti-drug antibodies | 224 | 226 | 450
  Week 12: number analyzed (Participants) | 226 | 226 | 452
  Week 12: Positive anti-drug antibodies | 1 | 2 | 3
  Week 12: Negative anti-drug antibodies | 225 | 224 | 449
  Week 24: number analyzed (Participants) | 225 | 225 | 450
  Week 24: Positive anti-drug antibodies | 6 | 6 | 12
  Week 24: Negative anti-drug antibodies | 219 | 219 | 438
  Week 48: number analyzed (Participants) | 229 | 225 | 454
  Week 48: Positive anti-drug antibodies | 9 | 12 | 21
  Week 48: Negative anti-drug antibodies | 220 | 213 | 433

17. Secondary Outcome: Anti-drug Antibodies Pre- and Post-first Dosing
Description: Number and percentage of patients with detection of anti-drug antibodies (ADAs) pre-first dosing and post-first dosing (combination of all ADA assessments after first injection of study medication).
Time Frame: Baseline and up to Week 48
Population: SAF
Measure: Count of Participants; unit: Participants
Arm/Group | FYB201 | Lucentis | Total
Number analyzed (Participants) | 238 | 239 | 477
Participants
  Pre-first dosing: number analyzed (Participants) | 232 | 236 | 468
  Pre-first dosing: Positive anti-drug antibodies | 0 | 5 | 5
  Pre-first dosing: Negative anti-drug antibodies | 232 | 231 | 463
  Post-first dosing: number analyzed (Participants) | 237 | 238 | 475
  Post-first dosing: Positive anti-drug antibodies | 14 | 14 | 28
  Post-first dosing: Negative anti-drug antibodies | 223 | 224 | 447

ADVERSE EVENTS:
Time Frame: From first treatment up to Week 48
Description: All Adverse Events are reported in this record from First Patient First Treatment until Last Patient Last Visit. SAF
Arm/Group | FYB201 | Lucentis
All-Cause Mortality (participants affected / at risk) | 2/238 | 1/239
Serious Adverse Events (participants affected / at risk) | 19/238 | 32/239
Other Adverse Events (participants affected / at risk) | 149/238 | 161/239
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FYB201 (N=238) | Lucentis (N=239)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (4) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 2 (2)
Iridocyclitis (Eye disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Endophthalmitis (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Catheterisation cardiac (Investigations) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Transient global amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Hydroureter (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary bladder polyp (Renal and urinary disorders) | 0 (0) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FYB201 (N=238) | Lucentis (N=239)
Cataract (Eye disorders) | 1 (1) | 10 (13)
Choroidal neovascularisation (Eye disorders) | 6 (6) | 4 (4)
Conjunctival haemorrhage (Eye disorders) | 14 (24) | 19 (30)
Conjunctival hyperaemia (Eye disorders) | 4 (4) | 6 (6)
Eye pain (Eye disorders) | 9 (14) | 6 (8)
Lacrimation increased (Eye disorders) | 9 (11) | 2 (2)
Neovascular age-related macular degeneration (Eye disorders) | 19 (19) | 22 (24)
Punctate keratitis (Eye disorders) | 8 (15) | 12 (25)
Retinal haemorrhage (Eye disorders) | 7 (9) | 3 (3)
Retinal pigment epithelial tear (Eye disorders) | 2 (2) | 6 (6)
Visual acuity reduced (Eye disorders) | 6 (6) | 11 (13)
Vitreous detachment (Eye disorders) | 6 (7) | 4 (4)
Vitreous floaters (Eye disorders) | 3 (3) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 5 (5)
Pain (General disorders) | 5 (9) | 2 (2)
Bronchitis (Infections and infestations) | 8 (8) | 5 (5)
Conjunctivitis (Infections and infestations) | 9 (10) | 2 (2)
Influenza (Infections and infestations) | 5 (7) | 2 (2)
Nasopharyngitis (Infections and infestations) | 12 (15) | 16 (17)
Upper respiratory tract infection (Infections and infestations) | 8 (10) | 6 (7)
Urinary tract infection (Infections and infestations) | 3 (3) | 6 (6)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 5 (5)
Blood urea increased (Investigations) | 4 (4) | 5 (5)
C-reactive protein increased (Investigations) | 10 (11) | 5 (5)
Intraocular pressure increased (Investigations) | 11 (20) | 12 (15)
Visual acuity tests abnormal (Investigations) | 4 (4) | 5 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 8 (8)
Dizziness (Nervous system disorders) | 1 (1) | 5 (5)
Headache (Nervous system disorders) | 4 (5) | 8 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 5 (5)
Hypertension (Vascular disorders) | 3 (6) | 14 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-08-29): https://cdn.clinicaltrials.gov/large-docs/78/NCT02611778/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-16): https://cdn.clinicaltrials.gov/large-docs/78/NCT02611778/SAP_001.pdf